CLINICAL TRIAL: NCT03608943
Title: Hydrocortisone Versus Prednisolone for Treatment of Adrenal Insufficiency Disease (HYPER-AID Study)
Brief Title: Hydrocortisone Vs Prednisolone in AI (HYPER-AID)
Acronym: HYPER-AID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 18HH4457; 234243 (Other: IRAS)
Record Dates: First submitted 2018-06-18; First posted 2018-08-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Adrenal Insufficiency
Keywords: glucocorticoids; prednisolone; hydrocortisone
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adrenal insufficiency: Individuals who are in the process of changing their treatment from:
  1. hydrocortisone to prednisolone or;
  2. prednisolone to hydrocortisone
  Interventions: Other: There is no specific intervention other than an individual changing their treatment as part of their usual care

INTERVENTIONS:
Other: There is no specific intervention other than an individual changing their treatment as part of their usual care — There is no specific intervention other than an individual changing their treatment as part of their usual care

SUMMARY:
This study is designed to collect data on individuals with adrenal insufficiency who are changing treatments from hydrocortisone to prednisolone, or vice versa. It will compare anthropometric, biochemical and subjective health outcomes between both treatments.

DETAILED DESCRIPTION:
In the UK, oral immediate release hydrocortisone divided in three doses daily has been the traditional treatment. The most common regimen in clinical practice uses doses of 10 mg on waking, 5 mg at lunch time and 5 mg in the afternoon. Once daily prednisolone is another regimen in clinical use and now prescribed at less than 5mg daily. It has a longer duration of action and a smoother pharmacokinetic profile compared to hydrocortisone. Moreover, prednisolone is much more cost-effective than hydrocortisone with 5mg tablets. Prednisolone is less commonly used due to perceived concerns regarding loss of bone mineral density leading to osteoporosis, increased insulin resistance leading to steroid induced diabetes, and rises in blood pressure and weight leading to increased cardiovascular risk. This belief is perhaps driven by the fact that most clinicians encounter prednisolone in the context of the treatment of asthma, rheumatoid arthritis etc. where far higher doses are employed. Where effects on bone health have been noted, they have been in association with higher doses of prednisolone (7.5mg) than those employed today (2-5mg).

Although conventionally prednisolone 5 mg is assumed to be bioequivalent to HC 20 mg (ratio 1:4), newer studies suggest that the ratio may be nearer 1:6-8 i.e. lower doses can be used.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 85 years
* Male or female
* Diagnosed with adrenal insufficiency (AI) for over 6 months according to standard diagnostic criteria
* Established on stable hydrocortisone or prednisolone replacement, dose not altered for at least 4 months
* Individuals taking other hormone replacements are accepted providing that their replacement doses have not altered for at least 3 months;
* Individuals who are able and willing to give written informed consent to participate in the study

Exclusion Criteria:

* Individuals who are unable to give informed consent
* Pregnancy (determined by patients self-reporting pregnancy status)
* Patients using the combined oral contraceptive pill

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with either primary or secondary adrenal insufficiency who are currently receiving glucocorticoid replacement therapy with hydrocortisone or prednisolone.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
P1NP | Minimum 4 months of stable treatment
  measurement of bone turnover markers: P1NP,
NTX | Minimum 4 months of stable treatment
  measurement of bone turnover markers: NTX

SECONDARY OUTCOMES:
Heart rate | Minimum 4 months of stable treatment
  recording observations- heart rate
Blood pressure | Minimum 4 months of stable treatment
  recording observations- blood pressure
Waist-hip circumference | Minimum 4 months of stable treatment
  recording observations- waist-hip circumference ratios
Lipid profile (Total cholesterol, HDL, LDL and triglycerides) | Minimum 4 months of stable treatment
  measuring biochemical indicators of cardiovascular risk: total cholesterol, HDL, LDL and triglycerides
High sensitivity CRP | Minimum 4 months of stable treatment
  measuring biochemical indicators of cardiovascular risk: high sensitivity CRP
Glucose | Minimum 4 months of stable treatment
  assessed by measuring glucose
HbA1c | Minimum 4 months of stable treatment
  assessed by measuring HBA1c
Frequency and severity of steroid replacement related symptoms | Minimum 4 months of stable treatment
  assessed by reporting of symptoms of steroid deficiency, their frequency and severity stratified by the patient's current replacement regimen. Symptoms include nausea, lethargy, muscle pain, headaches etc.)
Efficacy of replacement and wellbeing | Minimum 4 months of stable treatment
  assessed using subjective health questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Karim Meeran, MBBS BSc MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share individual data with other researchers